CLINICAL TRIAL: NCT06507267
Title: Pain and Clinical Reflections in Pelvic Congestion Syndrome,
Brief Title: Pain and Clinical Reflections in Pelvic Congestion Syndrome
Status: Recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: altunibrahim
Record Dates: First submitted 2024-04-24; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Pain, Chronic Primary
Keywords: Pelvic Congestion Syndrome, Pain,chronic pelvic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pain and Clinical Reflections in Pelvic Congestion Syndrome
  Interventions: Other: Pain and Clinical Reflections in Pelvic Congestion Syndrome

INTERVENTIONS:
Other: Pain and Clinical Reflections in Pelvic Congestion Syndrome — Pain and Clinical Reflections in Pelvic Congestion Syndrome

SUMMARY:
Pelvic congestion syndrome (PKS) occurs as a result of dysfunction of the veins in the pelvic area. It is currently called pelvic venous disease. This definition also includes some diseases of the pelvic region such as May-Thurner and Nutcracker syndrome. Dilatation and reflux are usually observed in the para-uterine or ovarian veins. PCS is one of the important causes of chronic pelvic pain (CPA). Pain in PCS is unrelated to the menstrual cycle. PCS is frequently seen in multiparous women in the reproductive period. Pregnancy worsens the clinical condition of patients with PCS due to mechanical pressure on the pelvic region vessels in pregnant women. Although the underlying cause of PCS is thought to be hormonal factors related to progesterone and estrogen, its etiology has not been fully elucidated and is thought to be multifactorial.GnRH analogues and medroxyprogesterone, which have side effects such as menstrual irregularity, osteoporosis and weight gain, were previously used in the medical treatment of PCS. Combined oral hormonal contraceptives, vasoactive flavonoid fraction drugs, nonsteroidal anti-inflammatory (NSAID) drugs for pain relief, Gabapentin, and Amiltriptyline are still used in the treatment of PCS. In the past, traditional hysterectomy and oophorectomy were performed surgically. Laparoscopic ovarian vein ligation has been performed since the early 2000s, but its popularity has decreased due to potential complications such as retroperitoneal hematoma, ureteral injury, and thrombosis. Endovascular intervention is more preferred today due to its low complications and high success in treatment.

DETAILED DESCRIPTION:
The study will be conducted by retrospectively scanning the files of patients diagnosed with pelvic congestion syndrome who underwent endovascular procedures with the plug method between January 2022 and March 2024 in the Cardiovascular Surgery Department of Kanuni Sultan Süleyman Training and Research Hospital. From the patients' files, age, body mass index (BMI), painful areas and painful side, medical treatments, comorbidities, onset of pain and application time for endovascular intervention, symptoms accompanying pain (feeling of heaviness in the perineum, swelling in the labia majora, dysuria, hematuria, dyspareunia) were obtained. , Postcoital pain, Dysmenorrhea, frequent urination) The position in which the pain increases, the branches consulted before endovascular intervention, and the Numerical Rating Scale-11 (NRS-11) score in the first and third months before and after the endovascular procedure for pain evaluation will be recorded on the patient follow-up form.

Numeric Rating Scale-11 (NRS-11) is an 11-point numerical scale in which patients can evaluate their pain between 0 (no pain) and 10 (the most severe pain they have ever felt in their life).

NRS-11 will be checked 3 times: before treatment, 1st month and 3rd month after treatment.

5. The number of patients and volunteers to be included in the research, their qualifications and the reason for selection (age ranges, gender, etc.).

The study was conducted in the Cardiovascular Surgery Department of Kanuni Sultan Süleyman Training and Research Hospital, from female patients between the ages of 18-50, who had abdominopelvic pain for more than 6 months, with clinical, physical examination and symptoms, and >6 mm in pelvic veins on transvaginal or transabdominal ultrasonography. It is planned to include 54 patients with over-dilatation.

ELIGIBILITY:
Inclusion Criteria:

* It is planned to include 54 female patients between the ages of 18-50,
* who have abdominopelvic pain for more than 6 months
* who have >6 mm dilatation in the pelvic veins on transvaginal or transabdominal ultrasonography along with clinical, physical examination and symptoms.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Exclusion Criteria:
  * In terms of gynecology, patients with leiomyoma, pelvic inflammatory disease,
  * endometriosis, postoperative adhesion,
  * patients who have undergone urological and gynecological surgery,
  * patients with chronic renal failure,
  * known allergies to the drugs used during the procedure,
  * patients with abdominopelvic trauma, malignancy or its history,
  * patients with a history of radiotherapy chemotherapy,
  * patients with known neuropsychiatric disorders.
  * Patients with disease,
  * pregnant women,
  * breastfeeding women,
  * fibromyalgia,
  * known lumbar disc herniation,
  * scoliosis,
  * facet syndrome,
  * sacroiliac dysfunction,
  * and patients with genitourinary and gastrointestinal diseases will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
onset of pain and application time for endovascular intervention, | 'four months'
  numerical rating scala - 11

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided